CLINICAL TRIAL: NCT01321177
Title: Recovery After an Initial Schizophrenia Episode (RAISE): RAISE Early Treatment Program
Brief Title: An Integrated Program for the Treatment of First Episode of Psychosis
Acronym: RAISE ETP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: State University of New York - Downstate Medical Center (Other); University of North Carolina, Chapel Hill (Other); University of California, Los Angeles (Other); Dartmouth-Hitchcock Medical Center (Other); Research Foundation for Mental Hygiene, Inc. (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John Kane, Chairman, Psychiatry, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHSN271200900019C; HHSN271200900019C (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2011-01-27; First posted 2011-03-23 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Brief Psychotic Disorder; Psychotic Disorder NOS
Keywords: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Brief Psychotic Disorder; Psychotic Disorder NOS; First Episode
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated Treatment (Experimental): Integrated program of treatments and services delivered by a coordinated team of providers.
  Interventions: Behavioral: Integrated Treatment
- Community Care (Active Comparator): Standard mental health treatments and services offered at the local agency.
  Interventions: Behavioral: Community Care

INTERVENTIONS:
Behavioral: Integrated Treatment — Integrated program of treatments and services delivered by a coordinated team of providers that includes:
  * education about schizophrenia and its treatment for the participants and their family members
  * medication for symptoms and preventing relapse that uses a computerized decision support system
  * strategies for managing the illness and building personal resilience
  * help getting back to school or work using a supported employment/education model
  Arms: Integrated Treatment
Behavioral: Community Care — Standard mental health treatments and services offered at the local agency that may include :
  * medication for symptoms and preventing relapse
  * psychosocial therapy which may include a range of behavioral treatments and supportive services
  * Case management
  Arms: Community Care

SUMMARY:
The purpose of this study is to determine how services should be provided to reduce symptoms and improve life functioning for adolescents and adults who have been recently diagnosed with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a major mental illness characterized by psychosis, negative symptoms (e.g., apathy, social withdrawal, anhedonia), and cognitive impairment. Depression and substance abuse commonly co-occur. These individuals have impaired functioning in the areas of work, school, parenting, self-care, independent living, interpersonal relationships, and leisure time. Among adult psychiatric disorders, schizophrenia is the most disabling, and its treatment accounts for a disproportionate share of mental health services.

This study is part of the National Institute of Mental Health's Recovery After an Initial Schizophrenia Episode (RAISE) Project. The RAISE Project seeks to fundamentally change the trajectory and prognosis of schizophrenia through coordinated and aggressive treatment in the earliest stages of illness. This study, the RAISE Early Treatment Program (ETP), is one of the two independent research studies that NIMH has funded to conduct the NIMH RAISE Project. ETP is being supported in whole or in part with Federal funds from the American Recovery and Reinvestment Act of 2009 and the NIMH, National Institutes of Health, Department of Health and Human Services.

The ETP study aims to compare two early treatment interventions for adolescents and adults experiencing a first episode of psychosis. The clinical centers have been randomly allocated to offer one of the two treatment programs. Both treatment interventions are designed to provide a person with treatment soon after he or she experiences the early signs of schizophrenia. Participants will be offered mental health services such as medication and psychosocial therapy. These strategies are all aimed at promoting symptom reduction and improving life functioning. Participation in this study will last between 2 and 3 years. All participants will first undergo an initial videoconference interview to confirm a diagnosis of schizophrenia, schizoaffective disorder, psychosis NOS, brief psychotic disorder, or schizophreniform disorder. Eligible participants will then be offered mental health services.

In addition to the mental health services, participants will participate in a series of research interviews. Participants will be interviewed every 3 months for the first 6 months and then every 6 months for up to 3 years. At the research visit, participants will complete an interview about their symptoms and general quality of life, complete questions about experiences with their illness, their vital signs will be measured, and a blood draw will be collected. At the initial, 12 and 24 month visits, participants will also complete a brief test that assesses skills such as memory, attention and problem solving. Participants will also have monthly telephone interviews about their illness and services that they have received.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SCID DSM-IV clinical diagnosis by trained remote clinical assessor of:

  * schizophrenia, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, psychotic disorder NOS
* Any duration of untreated psychosis
* Any ethnicity
* Ability to participate in research assessments in English
* Ability to provide fully informed consent (assent for those under age 18)

Exclusion Criteria:

* Inability to understand what research participation entails or correctly answer the questions about research participation that are part of the Study Information Review and provide fully informed consent
* More than 4 months of prior cumulative treatment with antipsychotic medications
* Diagnosis of bipolar disorder, psychotic depression or substance-induced psychotic disorder
* Current psychotic disorder due to a general medical condition
* Current neurological disorders that would affect diagnosis or prognosis. These would include, but are not limited to seizure disorders, dementing or degenerative disorders, lesions or substantial congenital abnormalities. In most cases, disorders such as headache disorders would not require protocol exclusion
* Clinically significant head trauma
* Any other serious medical condition that in the opinion of the investigator would seriously impair functioning making the patient unsuitable for the trial

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 404 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kane, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (33):
- United States (33):
  - San Fernando Mental Health Center, San Fernando, California
  - Santa ClaritaMental Health Center, Santa Clarita, California
  - Mental Health Center of Denver, Denver, Colorado
  - United Services Inc., Willimantic, Connecticut
  - Henderson Mental Health Center, Fort Lauderdale, Florida
  - Life management Center of Northwest Florida, Panama City, Florida
  - Central Fulton Community Mental Health Center, Atlanta, Georgia
  - Cobb County Community Services Board, Austell, Georgia
  - Park Center, Fort Wayne, Indiana
  - Community Mental Health Center, Inc., Lawrenceburg, Indiana
  - Eyerly Ball, Des Moines, Iowa
  - Terrebonne Mental Health Center, Houma, Louisiana
  - River Parish Mental Health Center, Laplace, Louisiana
  - Catholic Social Services of Washtenaw County (CSSW), Ann Arbor, Michigan
  - Touchstone Innovare, Grand Rapids, Michigan
  - Clinton-Eaton-Ingham Community Mental Health Authority, Lansing, Michigan
  - Human Development Center, Duluth, Minnesota
  - North Point Health and Wellness, Minneapolis, Minnesota
  - Pine Belt Mental Health Clinic, Hattiesburg, Mississippi
  - Burrell Behavioral Health, Columbia, Missouri
  - UMKC School of Pharmacy, Kansas City, Missouri
  - Burrell Behavioral Health, Springfield, Missouri
  - Community Alternatives, St Louis, Missouri
  - Community Mental Health Center of Lancaster County, Lincoln, Nebraska
  - The Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Greater Nashua Mental Health Center @ Community Council, Nashua, New Hampshire
  - Saint Clare's Hospital, Denville, New Jersey
  - University of New Mexico Department of Psychiatry UNM Health Sciences Center, Albuquerque, New Mexico
  - PeaceHealth Oregon/Lane County Behavioral Health Services, Eugene, Oregon
  - Lehigh Valley Hospital Mental Health Clinic, Allentown, Pennsylvania
  - South Shore Mental Health Center, Charlestown, Rhode Island
  - The Providence Center, Providence, Rhode Island
  - Howard Center, Burlington, Vermont

REFERENCES:
- [Derived] Mueser KT, Sussman RF, DeTore NR, Eberlin ES, McGurk SR. The impact of early intervention for first episode psychosis on cognitive functioning. Schizophr Res. 2023 Oct;260:132-139. doi: 10.1016/j.schres.2023.07.021. Epub 2023 Aug 30. PMID 37657279
- [Derived] Hong SI, Bennett D, Rosenheck RA. Gender differences in outcomes of early intervention services for first episode psychosis. Early Interv Psychiatry. 2023 Jul;17(7):715-723. doi: 10.1111/eip.13367. Epub 2023 Jan 9. PMID 36623822
- [Derived] Bornheimer LA, Cobia DJ, Li Verdugo J, Holzworth J, Smith MJ. Clinical insight and cognitive functioning as mediators in the relationships between symptoms of psychosis, depression, and suicide ideation in first-episode psychosis. J Psychiatr Res. 2022 Mar;147:85-93. doi: 10.1016/j.jpsychires.2022.01.006. Epub 2022 Jan 5. PMID 35026597
- [Derived] Bornheimer LA, Wojtalik JA, Li J, Cobia D, Smith MJ. Suicidal ideation in first-episode psychosis: Considerations for depression, positive symptoms, clinical insight, and cognition. Schizophr Res. 2021 Feb;228:298-304. doi: 10.1016/j.schres.2020.12.025. Epub 2021 Jan 23. PMID 33493778
- [Derived] Bornheimer LA, Tarrier N, Brinen AP, Li J, Dwyer M, Himle JA. Longitudinal predictors of stigma in first-episode psychosis: Mediating effects of depression. Early Interv Psychiatry. 2021 Apr;15(2):263-270. doi: 10.1111/eip.12935. Epub 2020 Feb 12. PMID 32052566
- [Derived] Robinson DG, Schooler NR, Rosenheck RA, Lin H, Sint KJ, Marcy P, Kane JM. Predictors of Hospitalization of Individuals With First-Episode Psychosis: Data From a 2-Year Follow-Up of the RAISE-ETP. Psychiatr Serv. 2019 Jul 1;70(7):569-577. doi: 10.1176/appi.ps.201800511. Epub 2019 May 14. PMID 31084291
- [Derived] Nuttall AK, Thakkar KN, Luo X, Mueser KT, Glynn SM, Achtyes ED, Kane JM. Longitudinal associations of family burden and patient quality of life in the context of first-episode schizophrenia in the RAISE-ETP study. Psychiatry Res. 2019 Jun;276:60-68. doi: 10.1016/j.psychres.2019.04.016. Epub 2019 Apr 16. PMID 31026764
- [Derived] Mueser KT, Meyer-Kalos PS, Glynn SM, Lynde DW, Robinson DG, Gingerich S, Penn DL, Cather C, Gottlieb JD, Marcy P, Wiseman JL, Potretzke S, Brunette MF, Schooler NR, Addington J, Rosenheck RA, Estroff SE, Kane JM. Implementation and fidelity assessment of the NAVIGATE treatment program for first episode psychosis in a multi-site study. Schizophr Res. 2019 Feb;204:271-281. doi: 10.1016/j.schres.2018.08.015. Epub 2018 Aug 20. PMID 30139553
- [Derived] Bornheimer LA. Suicidal Ideation in First-Episode Psychosis (FEP): Examination of Symptoms of Depression and Psychosis Among Individuals in an Early Phase of Treatment. Suicide Life Threat Behav. 2019 Apr;49(2):423-431. doi: 10.1111/sltb.12440. Epub 2018 Feb 14. PMID 29444349
- [Derived] Robinson DG, Schooler NR, Correll CU, John M, Kurian BT, Marcy P, Miller AL, Pipes R, Trivedi MH, Kane JM. Psychopharmacological Treatment in the RAISE-ETP Study: Outcomes of a Manual and Computer Decision Support System Based Intervention. Am J Psychiatry. 2018 Feb 1;175(2):169-179. doi: 10.1176/appi.ajp.2017.16080919. Epub 2017 Sep 15. PMID 28945118
- [Derived] Rosenheck RA, Estroff SE, Sint K, Lin H, Mueser KT, Robinson DG, Schooler NR, Marcy P, Kane JM; RAISE-ETP Investigators. Incomes and Outcomes: Social Security Disability Benefits in First-Episode Psychosis. Am J Psychiatry. 2017 Sep 1;174(9):886-894. doi: 10.1176/appi.ajp.2017.16111273. Epub 2017 Apr 21. PMID 28427286
- [Derived] Kane JM, Robinson DG, Schooler NR, Mueser KT, Penn DL, Rosenheck RA, Addington J, Brunette MF, Correll CU, Estroff SE, Marcy P, Robinson J, Meyer-Kalos PS, Gottlieb JD, Glynn SM, Lynde DW, Pipes R, Kurian BT, Miller AL, Azrin ST, Goldstein AB, Severe JB, Lin H, Sint KJ, John M, Heinssen RK. Comprehensive Versus Usual Community Care for First-Episode Psychosis: 2-Year Outcomes From the NIMH RAISE Early Treatment Program. Am J Psychiatry. 2016 Apr 1;173(4):362-72. doi: 10.1176/appi.ajp.2015.15050632. Epub 2015 Oct 20. PMID 26481174
- [Derived] Kane JM, Schooler NR, Marcy P, Correll CU, Brunette MF, Mueser KT, Rosenheck RA, Addington J, Estroff SE, Robinson J, Penn DL, Robinson DG. The RAISE early treatment program for first-episode psychosis: background, rationale, and study design. J Clin Psychiatry. 2015 Mar;76(3):240-6. doi: 10.4088/JCP.14m09289. PMID 25830446
- [Derived] Robinson DG, Schooler NR, John M, Correll CU, Marcy P, Addington J, Brunette MF, Estroff SE, Mueser KT, Penn D, Robinson J, Rosenheck RA, Severe J, Goldstein A, Azrin S, Heinssen R, Kane JM. Prescription practices in the treatment of first-episode schizophrenia spectrum disorders: data from the national RAISE-ETP study. Am J Psychiatry. 2015 Mar 1;172(3):237-48. doi: 10.1176/appi.ajp.2014.13101355. Epub 2014 Dec 4. PMID 25727536

RESULTS

PARTICIPANT FLOW:
Groups:
- Integrated Treatment: Integrated program of treatments and services delivered by a coordinated team of providers.
  Integrated Treatment: Integrated program of treatments and services delivered by a coordinated team of providers that includes:
  * education about schizophrenia and its treatment for the participants and their family members
  * medication for symptoms and preventing relapse that uses a computerized decision support system
  * strategies for managing the illness and building personal resilience
  * help getting back to school or work using a supported employment/education model
- Community Care: Standard mental health treatments and services offered at the local agency.
  Community Care: Standard mental health treatments and services offered at the local agency that may include :
  * medication for symptoms and preventing relapse
  * psychosocial therapy which may include a range of behavioral treatments and supportive services
  * Case management
Period: Overall Study
Arm/Group | Integrated Treatment | Community Care
Started | 223 | 181
Completed | 147 | 84
Not Completed | 76 | 97

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Treatment | Community Care | Total
Number analyzed (Participants) | 223 | 181 | 404
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 11 | 23
  Between 18 and 65 years | 211 | 170 | 381
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (5.2) | 23.1 (4.9) | 23.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 120 | 293
  Male | 50 | 61 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 18 | 73
  Not Hispanic or Latino | 168 | 163 | 331
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 223 | 181 | 404

OUTCOME MEASURES:

1. Primary Outcome: Mean Heinrichs-Carpenter Quality of Life Scale Scores Over Time
Description: This scale measures psychosocial functioning and behavior in people with schizophrenia. The scale contains 21 items rated 0 (no or minimal functioning) to 6 (normal functioning). The results are reported as the total score with a range from 0 to 126. Higher scores indicate a better outcome.
Time Frame: Baseline, Month 6, month 12, month 18 and month 24
Population: Intent to treat population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Integrated Treatment | Community Care
Number analyzed (Participants) | 223 | 181
score on a scale
  Baseline | 51.25 (0.89) | 55.13 (0.89)
  6 month | 59.15 (1.0) | 60.08 (1.12)
  12 month | 62.42 (1.21) | 62.12 (1.40)
  18 months | 64.93 (1.41) | 63.7 (1.66)
  24 months | 67.05 (1.59) | 65.02 (1.88)
Statistical Analysis 1: Comparison: Integrated Treatment vs Community Care; Test type: Superiority; p = 0.0145, Regression, Linear

2. Secondary Outcome: Positive and Negative Syndrome Scale for Schizophrenia (PANSS) Total Score
Description: This measures the presence and severity of symptoms of schizophrenia. The scales contains 30 items rated 1 (absent) to 7 (extreme). The results are reported in total score with a range of 30 to 210. Higher scores indicate a worse outcome.
Time Frame: Measured at baseline, month 6, month 12, month 18, and month 24
Population: Intent to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Integrated Treatment | Community Care
Number analyzed (Participants) | 223 | 181
score on a scale
  Baseline | 77.54 (0.94) | 74.69 (1.05)
  Month 6 | 70.38 (1.05) | 69.70 (1.16)
  Month 12 | 67.41 (1.17) | 67.63 (1.32)
  Month 18 | 65.14 (1.29) | 66.04 (1.46)
  Month 24 | 63.22 (1.4) | 64.7 (1.6)

3. Secondary Outcome: Calgary Depression Scale
Description: This scale is designed to assess depression in people with schizophrenia. The scale contains 9 items rated 0 (absent) to 3 (severe). The total score is reported and a higher value indicates a worse outcome. Total scores can range from 0 to 27. The data is reported as the estimated mean of the total score.
Time Frame: Measured at baseline, month 6, month 12, month 18, and month 24
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Integrated Treatment | Community Care
Number analyzed (Participants) | 223 | 181
score on a scale
  Baseline | 4.71 (0.24) | 4.52 (0.24)
  Month 6 | 3.72 (0.20) | 3.93 (0.21)
  Month 12 | 3.31 (0.21) | 3.68 (0.24)
  Month 18 | 3.00 (0.22) | 3.49 (0.26)
  Month 24 | 2.73 (0.24) | 3.33 (0.29)

4. Secondary Outcome: Service Use Rating Form (SURF)
Description: Measures of treatment services used
Time Frame: Measured at baseline and then monthly for months 1 through 24; reported as the monthly mean
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Services received
Arm/Group | Integrated Treatment | Community Care
Number analyzed (Participants) | 223 | 181
Services received | 4.53 (5.07) | 3.67 (5.93)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected during this study. Serious Adverse Events (SAEs) were collected throughout the study period which is defined from the time that the informed consent document is signed until 30 days after the last study visit/session, up to 25 months. SAEs occurring more than 30 days after a participant is discontinued from the study will be reported only if the investigator believes that the event may have been caused by a protocol-related procedure.
Description: Serious Adverse Events (SAEs) are defined as events that result in Death, inpatient hospitalization, a life-threatening experience, medically significant event not requiring hospitalization, persistent or significant disability/capacity, congenital anomaly/birth defect. Suicide attempts will be reported as SAEs, regardless of whether or not they result in hospitalization.
Arm/Group | Integrated Treatment | Community Care
All-Cause Mortality (participants affected / at risk) | 1/223 | 0/181
Serious Adverse Events (participants affected / at risk) | 71/223 | 66/181
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Treatment (N=223) | Community Care (N=181)
Psychiatric Hospitalization/illness (Psychiatric disorders) | 67 (121) | 63 (134)
Medical hospitalization/illness (General disorders) | 7 (8) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No